CLINICAL TRIAL: NCT00452374
Title: A Phase I-II Study of Oxaliplatin, Fludarabine, Cytarabine and Rituximab in Patients With Richter's Transformation, Prolymphocytic Leukemia or Refractory/Relapsed B-Cell Chronic Lymphocytic Leukemia
Brief Title: Oxaliplatin, Fludarabine, Cytarabine and Rituximab in Richter's Syndrome, Refractory CLL and PLL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0373
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; Chronic Lymphocytic Leukemia; CLL; Prolymphocytic Leukemia; PLL; Richter's Transformation; High-grade non-Hodgkin's lymphoma; Hodgkin's disease; Acute leukemia; Small lymphocytic lymphoma; Oxaliplatin; Eloxatin; Fludarabine; Cytarabine; Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride; Rituximab; Rituxan
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Hodgkin Disease | interventions — Cytarabine; fludarabine; fludarabine phosphate; Oxaliplatin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxaliplatin, Fludarabine, Cytarabine + Rituximab (Experimental): Starting dose oxaliplatin 17.5mg/m^2/day intravenous (IV) for 4 days; Fludarabine 30 mg/m^2 IV and Cytarabine 1 g/m^2 IV for two days, + Rituximab 375 mg/m^2 IV on Day 3, Cycle 1 then Day 1 following cycles.
  Interventions: Drug: Cytarabine; Drug: Fludarabine; Drug: Oxaliplatin; Drug: Rituximab

INTERVENTIONS:
Drug: Cytarabine — 1 g/m^2 given IV for two days (Days 2 and 3).
  Other Names: Ara-C; Cytosar; DepoCyt; Cytosine arabinosine hydrochloride
Drug: Fludarabine — 30 mg/m^2 given IV for two days (Days 2 and 3).
  Other Names: Fludara; Fludarabine Phosphate
Drug: Oxaliplatin — Starting dose of 17.5 mg/m^2 IV for 4 days (Days 1 through 4).
  Other Names: Eloxatin
Drug: Rituximab — 375 mg/m^2 IV on Day 3 of the first cycle over 4-6 hours and on Day 1 on every cycle following.
  Other Names: Rituxan

SUMMARY:
Primary Objectives:

1. Determine the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of oxaliplatin in combination with fludarabine, Ara-C and rituximab in patients with Richter's transformation, prolymphocytic leukemia (PLL), or refractory/relapsed B-cell chronic lymphocytic leukemia (CLL).
2. Assess the complete response (CR) and partial response (PR) rate to combination therapy of oxaliplatin, fludarabine, Ara-C and rituximab in patients with Richter's transformation, PLL or refractory/relapsed B-cell CLL.
3. Determine the safety and toxicity profile of combination therapy of oxaliplatin, fludarabine, Ara-C and rituximab in patients with Richter's transformation, PLL or refractory/relapsed B-cell CLL.

Secondary Objectives:

1. Determine the duration of response, failure-free survival, and overall survival.
2. Determine the incidence of infections (bacterial, fungal, and viral) in patients with Richter's transformation, prolymphocytic leukemia or refractory/relapsed B-cell CLL treated with rituximab, oxaliplatin, fludarabine and Ara-C; monitor immune parameters such as T cell counts and immunoglobulin levels; and monitor Epstein-Barr virus (EBV) status.
3. Characterize the pharmacodynamics of oxaliplatin in leukemia cells with respect to total adduct formation, cross-link formation and excision deoxyribonucleic acid (DNA) responses. Compare these parameters in cells from the same patient after treatment with oxaliplatin in combination with fludarabine and Ara-C.

DETAILED DESCRIPTION:
Oxaliplatin, fludarabine, cytarabine and rituximab are anticancer drugs. Oxaliplatin is a platinum compound that has been shown to be effective in fighting other cancers. Oxaliplatin is a third generation platinum compound with higher activity and less toxicity in colon cancer and other tumors compared to other platinum compounds, such as cisplatin. Oxaliplatin has shown activity in patients with relapsed or refractory non-Hodgkin's lymphoma.

Before treatment starts, you will have a complete physical exam and routine blood tests (about 2 teaspoons). A bone marrow sample will be collected. To collect a bone marrow sample, an area of the hip or chest bone is numbed with anesthetic and a small amount of bone marrow is withdrawn through a large needle. Women who are able to have children must have a negative blood or urine pregnancy test.

This research study has two parts, a Phase I part and a Phase II part. You will receive at least 1 cycle of therapy.

Oxaliplatin will be given through a needle in your vein (called an IV) for 4 days (Days 1 through 4). Rituximab will be given through an IV on Day 3 of the first cycle and on Day 1 on every cycle after that. One day after the first dose of oxaliplatin and rituximab (Day 2), fludarabine and cytarabine will be given through an IV for two days (Days 2 and 3). Peg-filgrastim will be given subcutaneously (through a needle just under your skin) on Day 6. Other IV fluids such as saline will be given on all of the treatment days to keep you from being dehydrated, which means that the daily visit may take eight hours. The combination will be repeated once a cycle (every 28 days) for up to a total of 6 cycles.

During the Phase I and II phases of the study, researchers will be testing different dose levels of the study drug combination. Three patients will be enrolled at each dose level. Each time the dose level is raised, it will occur after each patient has been monitored for 28 days. Individual patients who do not experience serious drug-related side effects after the second cycle may receive the next higher dose level for the following treatment cycles.

Drugs will be given before each dose of rituximab to lower the risk of side effects. If side effects do occur during rituximab treatment, rituximab may have to be stopped until the side effects go away and then restarted. This may make your time in the outpatient area longer.

The first treatment cycle will be given at M. D. Anderson. Depending on your response to treatment, up to 5 more cycles can be performed either at M. D. Anderson or at home with your regular physician. After 3 cycles of treatment, you will be checked at M. D. Anderson to see if the disease is responding to treatment. If the disease is responding after 3 cycles of therapy, you may continue to receive therapy for up to 3 more cycles. If the disease is not responding, you will be taken off the study and your doctor will discuss other treatment options with you.

Once the best safe dose of the drug combination is found in the Phase I portion of the study, the next group of participants entering the study will take part in the Phase II portion of the study. The goal of this part of the study is to look at the effects of the drug combination in patients with refractory CLL, prolymphocytic leukemia or Richter's transformation. The dose level for the combination will be the one found in the Phase I part of the study.

The same dose levels for all four drugs will be used throughout the Phase II portion of the study, unless intolerable side effects occur. In that case, the dose may be lowered or the treatment may be stopped. You will be taken off study if the disease gets worse.

During each treatment cycle, you will have blood samples (about 1 teaspoon each) taken once every 1-2 weeks. Bone marrow biopsies will be done at the end of the 3rd and 6th chemotherapy cycles.

After your last cycle of treatment is completed, you will have blood drawn (about 2 teaspoons each) every 3 months for as long as you are in remission, for routine testing.

This is an investigational study. The FDA has authorized the use of these drugs for research only, when given for this purpose. All of these drugs are commercially available for other types of treatment. Oxaliplatin will be free of charge during the study. You and/or your insurance company will be responsible for the cost of the other drugs used in this study. Patients will be enrolled at M. D. Anderson, University of California, San Diego, or Dana-Farber Cancer Institute. Up to 52 patients will take part in this multicenter study. The estimated number of patients who will be treated at M. D. Anderson is up to 52.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed Richter's transformation, fludarabine-refractory chronic lymphocytic leukemia or prolymphocytic leukemia.
2. Patients must be 18 years of age or older.
3. Patients must have a performance status of 0-2 (Zubrod scale).
4. Patients must have adequate renal function (serum creatinine below or equal to 2mg/dL or creatinine clearance greater than 30mL/min), unless renal dysfunction is considered due to organ infiltration by disease.
5. Patients must have adequate hepatic function (bilirubin less than or equal to 2.0 mg/dl; Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) less than or equal to 3 times the upper limit of normal (ULN) for the reference lab unless considered due to leukemia or congenital hemolytic disorder (for bilirubin).
6. Female patients of childbearing potential (including those <1 year post-menopausal) and male patients must agree to use contraception.
7. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital.
8. Patients must have platelet counts greater or equal to 20,000, unless due to disease involvement, or autoimmune disorders.

Exclusion Criteria:

1. Untreated or uncontrolled life-threatening infection.
2. Oxaliplatin, fludarabine, cytarabine or rituximab intolerance.
3. Pregnancy or lactation.
4. Chemotherapy and/or radiation therapy within 4 weeks.
5. Medical condition, including mental illness or substance abuse, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-11; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Wierda, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - University of California-San Diego, La Jolla, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/15/04 to 4/24/07. All patients registered at the University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Oxaliplatin, Fludarabine, Cytarabine + Rituximab
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oxaliplatin, Fludarabine, Cytarabine + Rituximab
Number analyzed (Participants) | 48
Age Continuous [Median (Full Range); unit: years] | 61 [37 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 34
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) Oxaliplatin
Description: MTD defined as dose level at which 2/3 or 2/6 participants experience Dose Limiting Toxicity (DLT), where DLTs are any oxaliplatin-related ≥Grade 3 non-hematological toxicity involving a major organ system (brain, heart, kidney, liver, lung) in the National Cancer Institute (NCI) Version 3.0 toxicity scale.
Time Frame: From treatment onset to end of each cycle of treatment (every 21 days)
Population: Of the 48 study participants, 19 were enrolled in the Phase I MTD group and included in the MTD analysis.
Measure: Number; unit: mg/m^2
Arm/Group | Oxaliplatin, Fludarabine, Cytarabine + Rituximab
Number analyzed (Participants) | 19
mg/m^2 | 25

2. Secondary Outcome: Number of Participants With a Complete Response or Partial Response
Description: According to International Workshop Response Criteria for Non-Hodgkin's Lymphomas: Complete remission (CR) defined as > 30% lymphocytes in the bone marrow, recovery of blood counts and no clinical symptoms; and Partial remission (PR) defined as > 50% decrease of clinical symptoms from baseline and recovery from blood counts.
Time Frame: Evaluation every 3 cycles of treatment (28 days per cycle), approximately 90 days
Measure: Number; unit: Participants
Arm/Group | Oxaliplatin, Fludarabine, Cytarabine + Rituximab
Number analyzed (Participants) | 48
Participants
  Complete response (CR) | 12
  Partial response (PR) | 28

ADVERSE EVENTS:
Time Frame: 1 year, 9 months
Arm/Group | Oxaliplatin, Fludarabine, Cytarabine + Rituximab
Serious Adverse Events (participants affected / at risk) | 28/48
Other Adverse Events (participants affected / at risk) | 48/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin, Fludarabine, Cytarabine + Rituximab (N=48)
Infection (Infections and infestations) | 11 (12)
Neutropenic Fever (Infections and infestations) | 9 (11)
Dehydration (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 4 (4)
Fever (General disorders) | 5 (5)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Left Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Retinal Hemorrhage (Vascular disorders) | 1 (1)
Gastrointestinal Hemorrhage (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxaliplatin, Fludarabine, Cytarabine + Rituximab (N=48)
Neutropenia (Blood and lymphatic system disorders) | 48 (48)
Anemia (Blood and lymphatic system disorders) | 48 (48)
Thrombocytopenia (Blood and lymphatic system disorders) | 48 (48)
Fatigue (General disorders) | 20 (20)
Nausea (Gastrointestinal disorders) | 13 (13)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Constipation (Gastrointestinal disorders) | 5 (5)
Pain (General disorders) | 5 (5)
Anorexia (Gastrointestinal disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Neuropathy (Nervous system disorders) | 4 (4)
Dehydration (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes